CLINICAL TRIAL: NCT05454878
Title: A Cohort Study of Atrial Fibrillation Monitoring on Patients With Lymphoma After Chemotherapy by Applying Wearable Electrocardiogram
Brief Title: Atrial Fibrillation Monitoring on Patients With Lymphoma After Chemotherapy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Yun Dai Chen, professor, Chinese PLA General Hospital
Other Study IDs: LAF-20220523
Record Dates: First submitted 2022-07-07; First posted 2022-07-12 (Actual); Last update posted 2022-07-12 (Actual); Status verified 2022-06

CONDITIONS: Atrial Fibrillation
Keywords: lymphoma; chemotherapy; atrial fibrillation
MeSH Terms: conditions — Atrial Fibrillation; Lymphoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This prospective cohort study is to investigate the incidence of atrial fibrillation after chemotherapy by aplying wearable ECG recoder and the risk factors on patients with newly diagonsed lymphoma

DETAILED DESCRIPTION:
This prospective, single-centre, observational cohort study is disigned to enroll 100 newly diagnosed lymphoma patients who met the inclusion and exclusion criteria to monitor the onset of atrial fibrillation and other arrhythmias during chemotherapy by using wearable ECG recorder, and to evaluate the incidence of atrial fibrillation and related risk factors.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years old;
2. Concurrent chemotherapy on patients with new-onset lymphoma: chemotherapy regimens containing anthracyclines;
3. The subject voluntarily signed the informed consent.

Exclusion Criteria:

1. With heart failure, acute stroke or acute coronary syndrome within 3 months before admission
2. With Atrial fibrillation on admission
3. Patient after pacemaker surgery
4. With mental illness or mentally disabled
5. Patients that the investigator considers as unsuitable for this test

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The new-onset lymphoma patient who was scheduled for chemotherapy
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-07-15 (Estimated); Primary Completion 2023-07-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Incidence | 1 year after the first course of chemotherapy
  Incidence of atrial fibrillation after chemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Yundai Chen, MD, Principal Investigator — Chinese PLA General Hospital
Locations (1):
- General hospital of PLA, Beijing, Beijing Municipality, China